CLINICAL TRIAL: NCT04478006
Title: Driving Therapeutic Progress of Childhood Leukemia Through Advanced Translational Research With Immediate and Long-term Impact. Precision Medicine for Childhood Leukemia.
Brief Title: Advanced Translational Research on Childhood Leukemia
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Kathy Chan, Scientific Officer, Chinese University of Hong Kong
Other Study IDs: HKCH-REC-2020-012; PAED-2024-082 (Other: IRB Central)
Record Dates: First submitted 2020-07-14; First posted 2020-07-20 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Childhood Leukemia
MeSH Terms: interventions — RNA-Seq

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood or bone marraw
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Childhood Leukemia: Peripheral blood and bone marrow samples are collected for genetic analysis, invitro drug sensitivity test and animal experiment.
  Interventions: Genetic: RNA-seq; Genetic: whole exon sequencing; Other: Cytogenetics test

INTERVENTIONS:
Genetic: RNA-seq — Gene expression and fusion transcripts analysis
Genetic: whole exon sequencing — Genetic alternation analysis
Other: Cytogenetics test — Remission and relapse are monitored by cytogenetic analyses.

SUMMARY:
Prognosis of children with leukemia, the most common pediatric cancer, has improved markedly. Yet, relapse still occurs in 15-40% of patients with a probability of survival of <50%, which is unlikely to be boosted by intensification of standard chemotherapy due to overwhelming toxicity. The advent of effective and safe targeted therapies for high-risk cases is therefore imperative. This study constitutes two research projects aiming at driving therapeutic advances.

DETAILED DESCRIPTION:
The first part of the study aimed to investigate genomics and drug sensitivity profiling of childhood leukemia and its potential application for precision medicine.

The second part of the study aimed to develop novel antibody for treatment of childhood leukemia by animal model experiments.

Design:

Project 1: Whole-exome and RNA sequencing will be performed on children with leukemia (ALL, AML, MPAL, JMML, MDS) prospectively recruited in the Hong Kong Children's Hospital. Samples will be screened for their sensitivity to preselected, clinically accessible targeted agents in an ex vivo culture system. Results for the high-risk patients will be subjected to the tumor broad for evaluation.

Project 2: Fully human antibody candidates identified by phage display will be engineered into therapeutic forms, and assessed for efficacy and safety in patient-derived xenografts of relapsed/refractory B-ALL and in transgenic mice. The mechanisms of action will be identified by single-cell RNA sequencing.

Significance:

Implementation of functional genomics could identify leukemia patients who will benefit from targeted therapies and enable tailoring of precision medicine. The invented antibodies could be moved forward into clinical trials for salvaging high-risk pediatric B-ALL. Immediate and long-term impact on therapy of childhood leukemia is foreseen.

ELIGIBILITY:
List of inclusion criteria:

1. acute lymphoblastic leukemia (ALL) or
2. acute myeloid leukemia (AML) or

3 .mixed phenotype acute leukemia (MPAL) or

4. juvenile myelomonocytic leukemia (JMML) or

5. myelodysplastic syndromes (MDS) or

6. normal bone marrow donor

List of exclusion criteria:

1. This study will not recruit subjects who are unable to understand English or Chinese.
2. Patient or parent refusal

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children suspected or diagnosed with leukemia at presentation will be recruited for the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Genetic alterations of childhood leukemia | Baseline
  Association of mutation data with drug sensitivity profiles and disease-free survival /overall survival are analysed using standard statistical methods.
Gene expression profiles of childhood leukemia | Baseline
  Global transcriptome and fusion transcripts of leukemic blasts are identified by RNA-sequencing.
Drug sensitivity profiles | Baseline
  Drug sensitivity results of individual patient blasts-derived ex vivo culture are presented as IC50 and AUC values.
Antibody efficacy for treatment of childhood leukemia | Up to 1 year
  In vitro biochemical and biological assays and invivo leukemic patient-derived xenografts are used to characterize the efficacy and toxicity of the novel human anitbodies.

CONTACTS AND LOCATIONS:
Overall Officials: Kam Tong Leung, Ph. D., Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Hong Kong Children Hospital, Hong Kong, Hksar, China